CLINICAL TRIAL: NCT00000328
Title: Buprenorphine/Naloxone Treatment for Opioid Dependence-Experiment III
Brief Title: Buprenorphine/Naloxone Treatment for Opioid Dependence-Experiment III) - 3
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-11160-3; 1R01DA011160 (NIH); R01-11160-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Heroin Dependence; Opioid-Related Disorders
Keywords: drug dependence
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Opioid-Related Disorders

SUMMARY:
The purpose of this study is to compare the clinical efficacy of the buprenorphine/naloxone combination tablet to methadone for opioid maintenance treatment.

DETAILED DESCRIPTION:
S/A brief "Summary for the Public"

ELIGIBILITY:
Inclusion Criteria:

Individuals must be at least 18 years of age, currently opioid dependent and meet FDA criteria for narcotic maintenance treatment. Co-morbid substance abuse or dependence disorders may also be present. Individuals must be healthy despite drug dependency.

Exclusion Criteria:

Individuals with evidence of an active Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) Axis I psychiatric disorder (e.g. psychosis, manic-depressive illness, organic psychiatric disorders), significant medical illness (e.g. liver or cardiovascular disease) or pregnant female subjects are excluded from study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1997-07; Primary Completion 1997-08 (Actual); Study Completion 1997-08 (Actual)

PRIMARY OUTCOMES:
Drug use
Retention
Opioid agonist rating
Opioid antagonist rating
Compliance
Medication identification
Addiction Severity Index (ASI) Composite Score Rating

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Amass, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States